CLINICAL TRIAL: NCT02771223
Title: Quantification of Thrombocytes Number and Function in Patients Undergoing Prolonged Extracorporeal Circulation for Cardiac Surgery
Brief Title: Quantification of Thrombocytes Number and Function in Patients Undergoing Prolonged Extracorporeal Circulation
Acronym: CPB-PLT-FNCT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Dr. Amit Lehavi MD FANZCA, Director of Pediatric Anesthesia, Rambam Health Care Campus
Other Study IDs: 15-645
Record Dates: First submitted 2016-04-22; First posted 2016-05-13 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Coagulopathy
MeSH Terms: conditions — Hemostatic Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study group: patients scheduled for prolonged cardiac surgery (over 3 hours anticipated ECC time) with no known coagulation disorders

SUMMARY:
Prolonged extracorporeal circulation (ECC) for cardiac surgery results in coagulation abnormalities, most of which related to the direct, time dependent effect of the polymer tubing and the pump rollers on the thrombocytes. Significant evidence demonstrates the effect of the duration of cardiopulmonary bypass on thrombocytes number and function, as well as on postoperative coagulopathy

DETAILED DESCRIPTION:
Quantification of the effect of ECC duration on blood coagulation and platelet number and function

* Observational study on 20 patients undergoing prolonged ECC
* Blood sampling every 30 minutes for platelet count, platelet adhesion markers and coagulation studies
* Blood test to be performed in Rambam Blood Bank Laboratory

ELIGIBILITY:
Inclusion Criteria:

* adults over 18 yo
* scheduled for prolonged cardiac surgery requiring ECC time over 3 hours

Exclusion Criteria:

* documented coagulopathy
* antiplatelet therapy other then aspirin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adults over 18 yo scheduled for prolonged cardiac surgery requiring ECC time over 3 hours,
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-04 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Change in Platelet function apoptosis markers | 1st sample - less than 10 minutes after induction of anesthesia, 2nd sample - less than 3 minutes after termination of CPB, 3rd sample - 10 minutes after protamine administration for heparin reversal, after termination of CPB
  Platelet apoptosis by annexin V (Flow cytometry)
Change in Platelet function activation markers | 1st sample - less than 10 minutes after induction of anesthesia, 2nd sample - less than 3 minutes after termination of CPB, 3rd sample - 10 minutes after protamine administration for heparin reversal, after termination of CPB
  Platelet activation by P-selectin (Flow cytometry)

SECONDARY OUTCOMES:
Change in platelet count over time | Every 30 minutes - starting less than 10 minutes after induction of anesthesia, and for 7 hours or until termination of CPB and protamine administration - whichever comes first

IPD SHARING:
Plan to Share IPD: No